CLINICAL TRIAL: NCT00392821
Title: Phase I/II Trial of Sorafenib (Nexavar) and RAD001 (Everolimus)in the Treatment of Patients With Advanced Clear Cell Renal Cell Carcinoma
Brief Title: Dosing and Effectiveness Study of Sorafenib and RAD001 in the Treatment of Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 44; CRAD001C2480
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Sorafenib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 and Sorafenib (Experimental): RAD001 and Sorafenib
  Interventions: Drug: Sorafenib; Drug: RAD001

INTERVENTIONS:
Drug: Sorafenib — Sorafenib
  Other Names: Nexavar
Drug: RAD001 — RAD001
  Other Names: Everolimus, Zortress, Certican

SUMMARY:
This study is being done in 2 parts. The first part is to determine the dose of RAD001 that should be used in combination with sorafenib. The second part is using the above determined dose of RAD001 in combination with sorafenib to see how effective these 2 drugs are against advanced kidney cancer.

Participants will be asked to keep a pill diary.

DETAILED DESCRIPTION:
The drugs used in this trial are called targeted drugs as they target specific activities that are carried out by cancer cells that make them grow and spread. Sorafenib is an approved drug for the treatment of advanced kidney cancer. RAD001 is an experimental drug that has been used in other research studies with other types of cancer. In this trial, the use of RAD001 and sorafenib together for the treatment of kidney cancer is experimental. In the Phase I portion of this study 13-16 patients will be treated with the same dose of sorafenib and different doses of RAD001. The purpose is to see what is a safe dose of RAD001 when combined with sorafenib in the treatment of kidney cancer. Once this dose of RAD001 is determined, about 65 more patients will be treated to see how effective this combination of drugs is against this kidney cancer.

Both of these drugs are taken by mouth. Sorafenib will be taken twice a day. RAD001 is taken by mouth weekly. Patients will be able to continue treatment as long as their disease does not worsen or side effects become intolerable.

ELIGIBILITY:
Inclusion Criteria:

* Clinically documented metastatic or unresectable locally recurrent clear cell renal carcinoma
* Previous removal of kidney except if the size of the tumor was less than 5 cm or there was extensive liver or bone metastasis
* May have had no prior chemotherapy or up to 1 prior treatment regimen with immunotherapy or chemotherapy
* Performance status of 0-1
* Measurable disease
* Adequate liver, renal, and bone marrow function
* Must be able to give written informed consent
* Women able to become pregnant must have a negative pregnancy test
* Must be 18 or over
* Must be able to swallow pills

Exclusion Criteria:

* Prior treatment with sorafenib or m-TOR inhibitors
* History of acute MI within the last 6 months
* Active brain metastasis or patients with meningeal metastases
* Prior treatment for another cancer in the last 5 years
* Prior bleeding problems; coughing up or vomiting blood
* Non-healing wounds, ulcer, or long bone fracture
* Chronic use of systemic steroids or immunosuppressive agents
* Uncontrolled hypertension

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hainsworth, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (11):
- United States (11):
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Cancer Research, Marietta, Georgia
  - Baptist Hospital East, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Research Medical Center, Kansas City, Missouri
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1: sorafenib 400 mg BID and everolimus 35 mg once weekly
- Phase 1 Dose Level -1: Sorafenib 200 mg PO BID, everolimus 35 mg PO once weekly
- Phase II: 200 mg PO BID and everolimus 35 mg PO once weekly
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level -1 | Phase II
Started | 3 | 6 | 69
Completed | 0 | 0 | 0
Not Completed | 3 | 6 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level -1 | Phase II | Total
Number analyzed (Participants) | 3 | 6 | 69 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 44 | 47
  >=65 years | 1 | 5 | 25 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 21 | 24
  Male | 2 | 4 | 48 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 52 | 61
  Unknown or Not Reported | 0 | 0 | 17 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 2 | 6 | 67 | 75
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 69 | 78

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of Patients Treated at MTD/Phase II Dose Level
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response Rate (ORR) = Percentage of Patients Who Experience an Objective Response (CR+ PR) to Treatment. In oncology, this outcome measure is reported for all patients treated at the same dose level and is not separated into Phase I and Phase II. The phase I and phase II results are not separated out as the timing of their enrollment (early in phase 1 or later phase II) is not relevant to the outcome measure.
Time Frame: 18 months
Population: Pts who received MTD dose also called Phase II dose (Sorafenib 200 mg PO BID, everolimus 35 mg). The 6 phase I pts and 69 phase II pts treated at this dose level are combined to evaluate the efficacy of the MTD/phase II dose. The Ph I and Ph II results are not separated out as the timing of their enrollment (early in Ph 1 or later Ph II) is not relevant to the outcome measure. 3 Ph I patients who were not treated at the MTD are excluded as this Outcome Measure is for MTD/Phase II dose level only
Measure: Number (95% Confidence Interval); unit: percentage of evaluable patients
Arm/Group | RAD001 and Sorafenib
Number analyzed (Participants) | 75
percentage of evaluable patients | 13 [7 to 23]

2. Secondary Outcome: Progression-Free Survival for Patients Treated at MTD/Phase II Dose Level
Description: Progression is Defined Using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% Increase in the Sum of the Longest Diameter of Target Lesions, or a Measurable Increase in a Non-target Lesion, or the Appearance of New Lesions. Progression-free survival was defined as the interval from the date of study entry until the date of tumor progression or death for the patients treated at the MTD/Phase II dose level. This outcome measure is reported for all patients treated at the same dose level and is not separated into Phase I and Phase II. The phase I and phase II results are not separated out as the timing of their enrollment (early in phase 1 or later phase II) is not relevant to the outcome measure.
Time Frame: 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | RAD001 and Sorafenib
Number analyzed (Participants) | 75
Months | 5.45 [3.9 to 7.6]

ADVERSE EVENTS:
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level -1 | Phase II
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 21/69
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level -1 (N=6) | Phase II (N=69)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CNS Ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage, GI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infection - lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney stones (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pain - back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain - chest (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pain - stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Stabilization of thoracic spine (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular - atherosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level -1 (N=6) | Phase II (N=69)
Acne (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2) | 1 (2)
Albumin (Investigations) | 2 (2) | 0 (0) | 4 (7)
Alkaline Phosphatase (Investigations) | 3 (19) | 1 (1) | 8 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (21) | 0 (0) | 9 (20)
Anemia (Blood and lymphatic system disorders) | 1 (6) | 1 (1) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (7) | 2 (3) | 25 (66)
AST, SGOT (Investigations) | 3 (11) | 1 (2) | 5 (9)
Bilirubin - abnormal (Investigations) | 2 (8) | 0 (0) | 1 (1)
Blisters (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 3 (8)
Bronchiospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
CNS ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (15) | 1 (1) | 11 (15)
Constitutional symptoms, Other (Temperature intolerance) (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (General disorders) | 3 (16) | 2 (6) | 15 (20)
Creatinine increased (Investigations) | 3 (7) | 2 (4) | 9 (26)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 2 (14) | 3 (4) | 37 (120)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 7 (21)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3) | 5 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (9) | 19 (64)
Edema: limb (General disorders) | 1 (3) | 1 (1) | 10 (20)
Edema: NOS (General disorders) | 2 (7) | 0 (0) | 2 (2)
Edema:headandneck (General disorders) | 0 (0) | 0 (0) | 5 (7)
Elevated BUN (Investigations) | 2 (2) | 1 (1) | 4 (9)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (35) | 5 (8) | 47 (192)
fever (General disorders) | 0 (0) | 1 (1) | 9 (14)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (15)
Hand-Foot Syndrome (Skin and subcutaneous tissue disorders) | 3 (29) | 2 (3) | 19 (57)
Headache (General disorders) | 0 (0) | 1 (1) | 15 (53)
Hematologic: ANC (Investigations) | 1 (4) | 0 (0) | 7 (11)
Hematologic: Hemoglobin (Investigations) | 3 (23) | 5 (7) | 19 (62)
Hematologic: Platelets (Investigations) | 2 (15) | 1 (1) | 23 (64)
Hematologic: WBC (Investigations) | 2 (5) | 0 (0) | 14 (43)
Hematuria (Investigations) | 2 (3) | 0 (0) | 4 (10)
Hemorrhage(nose) (General disorders) | 0 (0) | 0 (0) | 6 (8)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Hyperchloridemia (Investigations) | 2 (4) | 0 (0) | 1 (1)
Hypercholesterolemia (Investigations) | 2 (12) | 0 (0) | 9 (28)
Hyperglycemia (Investigations) | 2 (11) | 0 (0) | 11 (23)
Hyperkalemia (Investigations) | 2 (4) | 0 (0) | 6 (8)
Hyperlipidemia (Investigations) | 0 (0) | 1 (1) | 7 (19)
Hypermagnesemia (Investigations) | 1 (1) | 1 (1) | 1 (1)
Hypernatremia (Investigations) | 1 (5) | 0 (0) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 2 (17) | 0 (0) | 24 (68)
Hypertriglyceridemia (Investigations) | 1 (4) | 0 (0) | 6 (16)
hyperuricemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypochloridemia (Investigations) | 1 (3) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 1 (3) | 0 (0) | 0 (0)
Hypomagnesemia (Investigations) | 1 (3) | 0 (0) | 1 (2)
Hyponatremia (Investigations) | 0 (0) | 1 (1) | 5 (9)
Hypophosphatemia (Investigations) | 2 (7) | 0 (0) | 7 (13)
Increased Alanine transaminase, ALT, SGPT (Investigations) | 2 (6) | 0 (0) | 3 (4)
Infection (Eye) (Infections and infestations) | 1 (5) | 0 (0) | 0 (0)
Infection (joint) (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Infection(Sinus) (Infections and infestations) | 0 (0) | 2 (2) | 4 (5)
Infection(Urinary) (Infections and infestations) | 0 (0) | 1 (1) | 4 (6)
insomnia (Psychiatric disorders) | 1 (1) | 1 (3) | 10 (42)
International normalized ratio - abnormal (Investigations) | 1 (1) | 0 (0) | 1 (4)
Metabolic/Lab, Other (abnormal CO2 ) (Investigations) | 1 (1) | 0 (0) | 0 (0)
Metabolic/Lab, Other (abnormal HCT) (Investigations) | 3 (13) | 0 (0) | 1 (1)
Metabolic/Lab, Other (abnormal Ketones) (Investigations) | 1 (3) | 0 (0) | 0 (0)
Metabolic/Lab, Other (abnormal LDH) (Investigations) | 3 (10) | 0 (0) | 0 (0)
Metabolic/Lab, Other(LDH) (Investigations) | 0 (0) | 1 (1) | 3 (5)
Mood Alteration (Anxiety) (Nervous system disorders) | 0 (0) | 0 (0) | 6 (20)
Mood Alteration (Depression) (Nervous system disorders) | 1 (1) | 0 (0) | 5 (16)
Mucositis/stomatitis (Infections and infestations) | 0 (0) | 1 (2) | 13 (19)
Nausea (General disorders) | 3 (7) | 3 (7) | 36 (90)
Neuropathy (motor) (Nervous system disorders) | 1 (13) | 0 (0) | 2 (2)
Neuropathy (NOS) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
neuropathy (sensory) (Nervous system disorders) | 1 (12) | 0 (0) | 4 (4)
Ocular, Other (difficulty, L eye) (Eye disorders) | 1 (8) | 0 (0) | 0 (0)
Pain (abdomen) (General disorders) | 1 (2) | 0 (0) | 10 (17)
Pain (back) (General disorders) | 0 (0) | 0 (0) | 12 (20)
Pain (chest) (General disorders) | 1 (1) | 0 (0) | 8 (8)
Pain (flank) (General disorders) | 1 (1) | 0 (0) | 3 (4)
Pain (joint) (General disorders) | 2 (2) | 1 (1) | 19 (26)
Pain (muscle) (General disorders) | 1 (2) | 0 (0) | 9 (17)
Pain (neck) (General disorders) | 1 (1) | 0 (0) | 3 (3)
Pain (skin) (General disorders) | 1 (3) | 0 (0) | 3 (4)
Partial Thromboplastin Time (PTT) (Investigations) | 1 (5) | 0 (0) | 0 (0)
Phosphorous (Investigations) | 1 (4) | 0 (0) | 1 (1)
Proteinuria (Investigations) | 3 (27) | 3 (10) | 20 (68)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (6) | 3 (5) | 11 (30)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (16) | 2 (7) | 35 (106)
Rigors/chills (General disorders) | 2 (5) | 0 (0) | 4 (5)
Sensory Neuropathy (General disorders) | 0 (0) | 0 (0) | 4 (15)
Shingles (General disorders) | 1 (1) | 0 (0) | 1 (2)
Stomatitis (Infections and infestations) | 0 (0) | 0 (0) | 8 (12)
Sweating (General disorders) | 2 (23) | 0 (0) | 3 (14)
Taste alteration (General disorders) | 1 (1) | 1 (2) | 11 (32)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Voice changes (General disorders) | 1 (1) | 0 (0) | 3 (3)
Vomiting (General disorders) | 2 (2) | 2 (2) | 14 (33)
weekness (General disorders) | 1 (4) | 0 (0) | 6 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.